CLINICAL TRIAL: NCT02490748
Title: Phase III Study of Radiofrquency Ablation Combined With Cytokine-induced Killer Cells for the Patients With Cervical Cancer
Brief Title: Radiofrquency Ablation Combined With Cytokine-induced Killer Cells for the Patients With Cervical Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First People's Hospital of Changzhou (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cervical001
Record Dates: First submitted 2015-07-02; First posted 2015-07-07 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RFA alone (No Intervention): Patients undergo radiofrequency ablation alone.
- RFA+CIK (Experimental): Autologous cytokine-induced killer cells were transfer via venous one week after RFA Interventions
  Interventions: Procedure: Radiofrequency ablation; Biological: Cytokine-induced killer cells

INTERVENTIONS:
Procedure: Radiofrequency ablation — Radiofrequency ablation is performed percutaneously under CT/US guidance
  Other Names: RFA
  Arms: RFA+CIK
Biological: Cytokine-induced killer cells — The patients received autologous cytokine-induced killer cells transfusion one week after RFA treatment.
  Other Names: CIK
  Arms: RFA+CIK

SUMMARY:
The purpose of this study is to determine whether combining of radiofrequency ablation (RFA) and cytokine-induced killer cells (CIK) transfusion can prolong survival of patients with cervical cancer.

DETAILED DESCRIPTION:
The primary objective is to evaluate whether RFA followed by CIK transfusion can prolong survival of patients with cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* They were systematic reviews based on randomized controlled trials (rcts). They were phase II rcts comparing chemotherapy with other systemic therapy agents or with no further treatment for recurrent, metastatic, or persistent cervical cancer.

they reported at least one of these outcomes: complete or partial response rate, overall or progression-free survival rate, adverse effects, or healthrelated quality of life (rcts reporting on heterogeneous populations-for example, women at a range of disease stages-were included if results were given separately for patients with recurrent, metastatic, or persistent cervical cancer).

Exclusion Criteria:

* studies evaluating the role of radiotherapy administered with chemotherapy, or second- or subsequent-line therapy options.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07; Primary Completion 2038-06 (Estimated); Study Completion 2040-06 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | 1 year
  Recurrence-free survival (RFS) was defined as the time from the date of RFA to the date of recurrence or the date of the last follow-up.